CLINICAL TRIAL: NCT02067507
Title: Increasing Human Papillomavirus Vaccine Uptake in Low-Income, Ethnic Minority Adolescents in Los Angeles County
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Roshan Bastani, Professor of Health Policy and Management, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA154549-01A1 (NIH)
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Human Papilloma Virus Infection
Keywords: Human Papillomavirus; Immunization; Oncogenic viruses; Cervical Cancer; Health Disparities
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): LACDPH Site: CDC-developed small media in preferred language
  AltaMed Health Services Corporation Site: Usual care - Standing order for the HPV vaccine; required web-based training module for medical assistants and nurses containing basic information on HPV, the HPV vaccine, and standing order implementation
  Northeast Valley Health Corporation Site: Usual care
- Tailored education and referral (Experimental): LACDPH Site: Tailored education and referral intervention administered at LACDPH Site
  Interventions: Behavioral: Tailored education and referral
- Staff training and patient reminders (Experimental): Staff training and patient reminders administered at AltaMed Health Services Corporation Site
  Interventions: Behavioral: Staff training and patient reminders
- Clinic-level reminder systems (Experimental): Clinic-level reminders administered at Northeast Valley Health Corporation Site
  Interventions: Behavioral: Clinic-level reminder systems

INTERVENTIONS:
Behavioral: Tailored education and referral — LACDPH Site: 5-minute tailored educational messages and clinic referral for vaccine plus tailored small media
  Arms: Tailored education and referral
Behavioral: Staff training and patient reminders — AltaMed Health Services Corporation Site: (1) Health care provider training on the importance of HPV vaccination, strategies to appropriately frame the HPV vaccine conversation, and recommended processes and procedures for vaccine delivery; (2) Staff training on the importance of HPV vaccination, strategies to promote uptake of the vaccine, and recommended processes and procedures for vaccine delivery; (3) Patient reminders and provider cues for follow-up doses; and (4) Organizational strategies to improve processes for vaccine delivery, in addition to usual care activities
  Arms: Staff training and patient reminders
Behavioral: Clinic-level reminder systems — Northeast Valley Health Corporation Site: Three different clinic-level reminder systems, including a mailed letter, automated/robo telephone call, or text message reminder
  Arms: Clinic-level reminder systems

SUMMARY:
The primary aim of the project is to increase human papillomavirus (HPV) vaccine receipt rates among low-income, ethnic minority adolescents (girls and boys 11-17 years of age) in Los Angeles County. We will accomplish this goal by implementing and rigorously evaluating interventions in multiple venues that serve our target population, including the Los Angeles County Department of Public Health (LACDPH) and two large Federally Qualified Health Centers (FQHCs).

Our hypotheses are:

Primary hypothesis:

1. The intervention group will have a higher rate of HPV vaccine initiation at follow-up compared to the control group.

   Secondary hypothesis:
2. The intervention group will have higher vaccine completion rates (3 doses) at follow-up compared to the control group.

DETAILED DESCRIPTION:
The primary aim of the project is to increase HPV vaccine receipt rates among low-income, ethnic minority adolescents (girls and boys ages 9-17 years) in LA County. We will accomplish this goal by implementing and rigorously evaluating interventions in multiple venues that serve our target population, including the Los Angeles County Department of Public Health (LACDPH) and two large Federally Qualified Health Centers (FQHCs).

Our hypotheses are:

Primary hypothesis:

1. The intervention group will have a higher rate of HPV vaccine initiation at follow-up compared to the control group.

   Secondary hypothesis:
2. The intervention group will have higher vaccine completion rates (3 doses) at follow-up compared to the control group.

Recruitment Venue 1: Los Angeles County Department of Public Health. At the LACDPH, the multi-component intervention will be directed at caregivers of age-eligible adolescents (11-17 years) and include brief individually-tailored telephone education, referral to a clinic offering low cost/free vaccine, and a mailed brochure. The control group will receive usual care and a standard Centers for Disease Control and Prevention (CDC) HPV vaccine fact sheet.

Additional secondary hypotheses for this recruitment venue include:

1. The intervention group will have higher knowledge of HPV and the HPV vaccine than the control group.
2. The intervention will have a greater effect on the more acculturated than less acculturated participants (moderator effect).
3. The intervention will exert its effect on vaccine receipt by increasing knowledge and reducing barriers (mediator effects).

This recruitment venue will utilize a two-arm time-randomized (on-off) controlled design to assess the effect of a multi-component intervention targeting mothers and fathers, to increase HPV vaccine uptake among their adolescents (ages 11-17). Hotline users will be randomized into the intervention or control condition on an alternating (on/off) weekly schedule. Eligible participants will complete a baseline telephone interview. Immediately following the baseline interview, participants calling during intervention weeks will receive the individually-tailored multi-component intervention, including tailored education and clinic referral. A tailored print intervention will also be mailed to intervention participants. All participants will be re-contacted at 3 months and 9 months for telephone follow-up interviews. Control group participants will receive the intervention after the 9-month follow-up. Prior to study protocol implementation, about 25-50 individuals will be recruited to pre-test the baseline survey in different languages (English, Spanish, Chinese, Armenian) to ensure the baseline questionnaires are similar in content across languages and the questions are clear.

The study site will enroll men and women of diverse racial-ethnic backgrounds from the Office of Women's Health (OWH) women's health telephone hotline database. The database includes contact information about adult women LA County residents who telephoned a 1-800 hotline to receive information and referrals about women's health issues, including cervical cancer and cervical cancer screening. Male callers also use the hotline. The OWH has promoted the hotline through partnerships with over 300 community-based organizations. Recruitment of callers from the database will consist of operators calling women to invite them to be screened for study eligibility. Recruitment of new hotline callers will take place during their first contact with the hotline. Upon receiving an incoming call, operators will first respond to the caller's request using routine hotline protocols which include screening for income eligibility (<200% of poverty) for county services. Following this, operators invite the caller to be screened for study eligibility. Eligible participants will be asked to complete the baseline interview.

Callers will be randomized to the intervention or control condition on alternating weeks (on-off or time randomized design). This randomization scheme was selected in close consultation with OWH to ensure the integrity of the randomization process and minimize disruption of routine hotline operation. The telephone intervention will be delivered immediately following the baseline telephone interview to participants calling during intervention weeks. The intervention is based on the Health Behavior Framework and pilot study findings and incorporates individual-level tailoring. The three segments of the telephone intervention include: 1) basic information about the HPV vaccine; 2) individually-tailored information to address each participant's primary concerns regarding the vaccine; 3) individually-tailored referral to a local clinic where free/low cost vaccine is available.

Baseline interviews (10-15 mins) will be conducted immediately following the eligibility screener and the verbal informed consent, via a Computer Assisted Telephone Interviewing System. All eligible subjects who complete the baseline interview will receive brief (<10 mins) 3 and 9-month follow-up telephone interviews.

Following the 3-month interviews, half of intervention participants will receive a "booster" intervention wherein we will repeat the clinic referral procedure/language given during the intervention at baseline. Intervention participants will be randomized to the "booster" or no "booster" condition based on the order in which they completed the baseline survey.

Recruitment Venue 2: AltaMed Health Services Corporation. At AltaMed Health Services Corporation, the largest federally qualified health center in the nation, we will implement a multi-level intervention that includes patient (i.e., caregiver) and provider reminders, physician, nurse, and other staff training regarding the HPV vaccine and processes and procedures for its delivery. We will utilize a quasi-experimental study design to assess the effect of this multi-level intervention to increase HPV vaccine initiation and completion among adolescents (ages 9-17). Eight clinic sites that serve the majority of AltaMed's adolescent population will be matched based on the size of the adolescent population served and baseline HPV vaccination rates. We will randomly assign matched paired clinics to either the intervention (n=4) or usual care group (n=4).

Clinics assigned to the usual care condition will only receive: (1) the standing order for the HPV vaccine, which authorizes non-physician providers to assess adolescents' immunization eligibility and administer the HPV vaccine without a physician examination or order and (2) a required web-based training module for medical assistants and nurses containing basic information on HPV, the HPV vaccine, and standing order implementation.

In addition to usual care activities, intervention clinics will receive the following: (1) health care provider training on the importance of HPV vaccination and a strong provider recommendation, strategies to appropriately frame the HPV vaccine conversation, and recommended processes and procedures for vaccine delivery; (2) staff training on the importance of HPV vaccination, strategies to promote uptake of the vaccine, and recommended processes and procedures for vaccine delivery; (3) patient and provider reminders to promote completion of the three-dose vaccine series; and (4) organizational strategies to improve processes for vaccine delivery, in addition to usual care activities.

The intervention will be developed in close collaboration with administrative leadership and providers, who will provide input at each stage of the design, implementation, and evaluation process. A physician vaccine champion from the organization will assist with the development of and lead a one-hour, in-person provider presentation and discussion. For the staff training presentation, nurse managers will be convened regularly to discuss processes for HPV and general standing order implementation, strategies to optimize clinical workflow and increase follow-up, and development of back office staff training. Using a train-the-trainer approach, the nurse mangers will lead the approximate one-hour presentation and discussion at their respective clinics. They will also monitor process implementation through direct staff observation and quality reports and retrain staff as needed.

In addition to provider and staff trainings, organizational strategies at intervention sites will include implementation of standard practices for HPV vaccine delivery that complement existing clinical workflow. At intake, back office staff will check vaccination history at each visit, implement needed standing orders, inform caregivers of vaccines due, and notify the provider of vaccines ordered. During the provider encounter, providers will confirm recommended vaccinations and recommend the HPV vaccine as part of other routine vaccines. At check-out, back office staff will administer vaccines, schedule a visit for the second dose, and provide caregivers both a standard appointment card and an intervention site reminder magnet. A clinic provider vaccine champion will be identified to monitor implementation, adapt processes, and serve as a resource at intervention sites.

To estimate intervention effects, we will use data extracted from AltaMed's electronic medical record system to measure HPV vaccine initiation and completion rates among adolescents ages 9-17 at baseline and at regular intervals post intervention implementation. Patient, provider and clinic factors associated with vaccine receipt will also be examined.

Recruitment Venue 3: Northeast Valley Health Corporation. At Northeast Valley Health Corporation, another large federally qualified health center, we will implement and evaluate the effects of three different clinic-level reminder systems (mailed letter, automated/robo telephone call, text message) on HPV vaccine initiation and completion among adolescents (ages 12-13).

We will utilize a quasi-experimental study design. This FQHC comprises 8 sites that provide primary care for medically underserved adults and adolescents in LA County. We will select 6 clinics matched on baseline vaccine receipt rates and other clinic characteristics and randomly assign matched paired clinics to usual care or one of the three reminder system interventions: mailed letter, automated/robo telephone call, or text message. Eligible caregivers of adolescent boys and girls ages 12-13 who have received no doses or only one dose of the HPV vaccine will be identified through Northeast Valley's electronic medical record and population health management systems.

After identification of eligible patients (i.e. caregivers), the centralized call center will generate a standard letter and the automated/robocalls. A third-party vendor will send the text messages. The reminder content will be adapted from existing clinical message scripts and include a short message, which will be consistent across all modalities, on the importance of HPV vaccination and how to make an appointment. Reminder messages will be delivered in the patients' preferred language (either English or Spanish). The same reminder type (either letter, call, or text message) will be used on up to two occasions: once at baseline and a second time approximately one month after baseline for those who have not yet received the targeted vaccine dose. To monitor receipt of reminders, number of unaccepted telephone calls, returned letters, and stopped text messages will be monitored. Clinics assigned to the usual care condition will receive standard of care, which does not include any systematic reminders.

Similar to the AltaMed FQHC site, to estimate intervention effects, we will use data extracted from electronic medical records to measure HPV vaccine initiation and completion rates at baseline and at regular intervals post intervention implementation.

ELIGIBILITY:
Recruitment Venue 1 (LACDPH) Criteria:

Inclusion Criteria:

* Adult male or female
* Current or previous user of the Los Angeles County Office of Women's Health Hotline
* Speaks one of the hotline languages (English, Spanish, Korean, Mandarin, Cantonese, Armenian)
* Is the medical decision-maker for a male or female adolescent aged 11-17 in his or her home
* Adolescent has not started the HPV vaccine series
* Current resident of Los Angeles County

Exclusion Criteria:

* Younger than 18 or older than 70 years of age
* Not conversant in one of the hotline languages (English, Spanish, Korean, Mandarin, Cantonese, Armenian)
* Is not the medical decision-maker for an adolescent aged 11-17 in his or her home
* Adolescent has initiated the HPV vaccine series
* Not a current resident of Los Angeles County

Recruitment Venue 2 (AltaMed) Criteria:

Inclusion Criteria:

* Adolescent male or female (9-17 years)
* Has received at least one service at the FQHC in the past 2 years

Exclusion Criteria:

* Younger than 9 or older than 17 years of age
* Has not received any services at the FQHC in the past 2 years

Recruitment Venue 3 (NEVHC) Criteria:

Inclusion Criteria:

* Adolescent male or female (12-13 years)
* Has received at least one service at the FQHC in the past 2 years
* Has received no doses or 1 dose of the HPV vaccine

Exclusion Criteria:

* Younger than 12 or older than 13 years of age
* Has not received any services at the FQHC in the past 2 years
* Has completed the 3-dose HPV vaccine

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53414 (Actual)
Dates: Start 2012-06; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
HPV Vaccine Uptake | 3 months, 6 months
  The receipt of one or more doses of the HPV vaccine

SECONDARY OUTCOMES:
HPV Vaccine Series Completion | 9 months, 12 months
  Completion of the 3-dose HPV vaccine series

OTHER OUTCOMES:
Knowledge and Attitudes Regarding HPV Vaccination | 9 months
  Participants' knowledge of and attitudes regarding HPV, cervical cancer, and the HPV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Bastani, PhD, Principal Investigator — University of California, Los Angeles; Beth Glenn, PhD, Study Director — University of California, Los Angeles
Locations (2):
- United States (2):
  - Los Angeles County Department of Public Health, Alhambra, California
  - Northeast Valley Health Corporation, San Fernando, California

IPD SHARING:
Plan to Share IPD: No